CLINICAL TRIAL: NCT00470327
Title: A Study of the Natural Progression of Interstitial Lung Disease (ILD)
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: Idiopathic Pulmonary Fibrosis Clinical Research Network (Network); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 14163A; 1R21AI126031-01 (NIH)
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Interstitial Lung Diseases; Idiopathic Pulmonary Fibrosis; Sarcoidosis; Connective Tissue Disorder
Keywords: Interstitial lung diseases; idiopathic pulmonary fibrosis; Sarcoidosis; mRNA and cytokine expression
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis; Sarcoidosis; Connective Tissue Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We propose to acquire data and blood samples on all patients being cared for by the Interstitial Lung Disease (ILD) program. Additionally, we will collect data and blood samples from a control group for comparator purposes. In doing so, we will be able to describe the "phenotypic" expression of these diseases.

ELIGIBILITY:
Inclusion Criteria:

* Interstitial lung disease

Exclusion Criteria:

* Does not have Interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects cared for in the ILD (Interstitial Lung Disease)clinic
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2005-09 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Natural history of course of disease in patients with Interstitial lung disease (ILD) | Yearly
  We assess mortality roughly yearly but duration is unlimited

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Strek, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share coded data with no PHI